CLINICAL TRIAL: NCT03261401
Title: A Phase I, First-in-Human, Randomized, Double-Blind, Placebo-Controlled Trial of Single and Multiple Ascending Doses of M5717 to Assess the Safety, Tolerability and Pharmacokinetic Profile of Oral Doses, and to Assess the Antimalarial Activity of M5717 Against Plasmodium Falciparum in Healthy Male and Female Adult Subjects
Brief Title: First-in-Human Trial of Single Ascending Dose, Multiple Ascending Dose and Malaria Challenge Model in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS201618_0013; 203481/Z/16/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2017-08-18; First posted 2017-08-25 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Healthy Participants; M5717; Malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part A: Placebo (Pooled) (Placebo Comparator): Participants received capsules containing 50 milligram (mg) of placebo matched similar to M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose.
  Interventions: Drug: Placebo
- Part A: Cohort 1 SAD: M5717 50 mg (Experimental): Participants received single ascending dose (SAD) of 50 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 2 SAD: M5717 100 mg (Experimental): Participants received SAD of 100 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 3 SAD: M5717 200 mg (Experimental): Participants received SAD of 200 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 4 SAD: M5717 400 mg (Experimental): Participants received SAD of 400 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 5 SAD: M5717 600 mg (Experimental): Participants received SAD of 600 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 6 SAD: M5717 1000 mg (Experimental): Participants received SAD of 1000 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 7 SAD: M5717 1250 mg (Experimental): Participants in SAD received an oral dose of 1250 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 8 SAD: M5717 1800 mg (Experimental): Participants in SAD received an oral dose of 1800 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part A: Cohort 9 SAD: M5717 2100 mg (Experimental): Participants in SAD received an oral dose of 2100 mg M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part C: Challenge Cohort 2 M5717 150 mg (Experimental): Participants received single oral dose of 150 mg M5717 (eight days after the administration of intravenous malaria inoculum) on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part C: Challenge Cohort 1 M5717 400 mg (Experimental): Participants received single oral dose of 400 mg M5717 (eight days after the administration of intravenous malaria inoculum) on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717
- Part C: Challenge Cohort 3 M5717 800 mg (Experimental): Participants received single oral dose of 800 mg M5717 (eight days after the administration of intravenous malaria inoculum) on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
  Interventions: Drug: M5717

INTERVENTIONS:
Drug: M5717 — Participants received single ascending oral dose of M5717 after at least 8 hours of fasting together with water on Day 1, followed by a 4-hour post-dose fast
  Arms: Part A: Cohort 1 SAD: M5717 50 mg; Part A: Cohort 2 SAD: M5717 100 mg; Part A: Cohort 3 SAD: M5717 200 mg; Part A: Cohort 4 SAD: M5717 400 mg; Part A: Cohort 5 SAD: M5717 600 mg; Part A: Cohort 6 SAD: M5717 1000 mg; Part A: Cohort 7 SAD: M5717 1250 mg; Part A: Cohort 8 SAD: M5717 1800 mg; Part A: Cohort 9 SAD: M5717 2100 mg
Drug: Placebo — Participants received placebo matched to M5717
  Arms: Part A: Placebo (Pooled)
Drug: M5717 — Participants received single ascending oral dose of M5717 from Part A after at least 8 hours of fasting together with water on Day 1, followed by a 4-hour post-dose fast
  Arms: Part C: Challenge Cohort 1 M5717 400 mg; Part C: Challenge Cohort 2 M5717 150 mg; Part C: Challenge Cohort 3 M5717 800 mg

SUMMARY:
The primary purpose of this study was to investigate the safety and tolerability of M5717 and to characterize the Pharmacokinetics (PK) /Pharmacodynamic relationship between M5717 PK and parasite clearance in healthy participants following infection with Plasmodium falciparum.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women of non-childbearing potential, with total body weight greater than or equal to 50.0 kilogram and body mass index (BMI) between 19.0 kilogram per meter square(kg/m^2) and 29.9 kg/m^2.
* Healthy as assessed by the Investigator with no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the trial evaluation, procedures, or completion.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Participants with history or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological dermatological, connective tissue diseases or disorders.
* Participants with history of relevant drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other allergic reaction in general, which the Investigator considers may affect the safety of the participant and/or outcome of the trial.
* Participants who have any history of malaria.
* Participants who have participated in a previous malaria vaccine trial.
* Participants who have participated in a previous human malaria challenge trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Q-Pharm Pty Ltd, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- [Result] McCarthy JS, Yalkinoglu O, Odedra A, Webster R, Oeuvray C, Tappert A, Bezuidenhout D, Giddins MJ, Dhingra SK, Fidock DA, Marquart L, Webb L, Yin X, Khandelwal A, Bagchus WM. Safety, pharmacokinetics, and antimalarial activity of the novel plasmodium eukaryotic translation elongation factor 2 inhibitor M5717: a first-in-human, randomised, placebo-controlled, double-blind, single ascending dose study and volunteer infection study. Lancet Infect Dis. 2021 Dec;21(12):1713-1724. doi: 10.1016/S1473-3099(21)00252-8. Epub 2021 Oct 26. PMID 34715032
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201618_0013
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 3 parts: Part A, B and C. Part B of the study was optional and sponsor decided not to perform part B of the study. In each cohort of Part A, participants were randomized in a 6:2 ratio to receive M5717 or matching placebo.
Groups:
- Part A: Placebo (Pooled): Participants from each cohort of Part A received single oral dose of placebo matched with M5717 on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose.
- Part C: M5717 150 mg: Participants received single oral dose of 150 mg M5717 (eight days after the administration of intravenous malaria inoculum) on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
- Part C: M5717 400 mg: Participants received single oral dose of 400 mg M5717 (eight days after the administration of intravenous malaria inoculum) on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
- Part C: M5717 800 mg: Participants received single oral dose of 800 mg M5717 (eight days after the administration of intravenous malaria inoculum) on Day 1 after 8 hours fasting-period followed by a 4-hour post-dose fast.
Period: Overall Study
Arm/Group | Part A: Placebo (Pooled) | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Started | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 6 | 8 | 8
Completed | 17 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 1 | 6 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Unable To Attend Final Visit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received investigational medicinal product (M5717 or placebo for Part A; M5717 for Part C).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo (Pooled) | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg | Total
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 6 | 8 | 8 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 5
  Between 18 and 65 years | 17 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 6 | 1 | 5 | 6 | 8 | 83
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 6 | 8 | 8 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 12
  Not Hispanic or Latino | 16 | 5 | 5 | 6 | 5 | 5 | 4 | 5 | 5 | 1 | 5 | 6 | 8 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 6
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4
  White | 13 | 4 | 4 | 6 | 5 | 6 | 2 | 5 | 4 | 1 | 4 | 4 | 8 | 66
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation of Study Treatment
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered with study drug which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 55
Population: Safety Analysis Set included all participants who received investigational medicinal product (M5717 or placebo for Part A).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo (Pooled) | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Participants
  TEAEs | 13 | 6 | 5 | 3 | 4 | 3 | 4 | 5 | 6 | 1
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs Leading to Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part A: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Assessments
Description: Laboratory assessments included hematology, biochemistry, urinalysis, and coagulation. Number of participants with clinically significant change from baseline in laboratory parameters were reported. Clinical significance was decided by the investigator.
Time Frame: Baseline up to Day 55
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo (Pooled) | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Clinically Significant Changes From Baseline in 12-lead Electrocardiograms (ECGs) Findings
Description: The 12-lead ECGs were recorded after the participants had rested for at least 5 minutes in supine position. Number of participants with clinically significant change from baseline in ECGs was reported. Clinical significance was decided by the investigator.
Time Frame: Baseline up to Day 55
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo (Pooled) | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate. Number of participants with clinically significant change from baseline in vital signs was reported. Clinical significance was decided by the investigator.
Time Frame: Baseline up to Day 55
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo (Pooled) | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Part C: Parasite Reduction Ratio (PRR) Assessed Through Quantitative Polymerase Chain Reaction (qPCR) Analysis
Description: The parasite reduction ratio (PRR) of asexual parasites based on quantitative polymerase chain reaction (qPCR) after administration of M5717 is a mathematical representation of the ratio of the parasite density between drug administration and for a defined period of time. The PRR for asexual forms was estimated using the slope of the optimal fit of the log-linear relationship of the parasitemia decay; ie, the time point where steady exponential decay in parasitemia occurs which may happen after a lag-phase. Lag phase is defined as an initial period after dosing that precedes a steady exponential decline in the parasite count. It was observed that the decline of parasitemia had a biphasic profile, with the first phase, followed by a second phase (the main clearance phase).
Time Frame: Day 1 to Day 22
Population: Pharmacodynamic (PD) analysis set included all participants who received M5717, had no clinically important protocol deviations or important events affecting PD and provided at least one (measurable) post-dose PD data. Here 'Number of Participants Analyzed' =number of participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 6 | 7
Ratio
  First Phase | 1.15 [0.59 to 2.25] | 1.73 [1.27 to 2.37] | 3.86 [2.9 to 5.13]
  Second Phase | 12892 [3858 to 43081] | 5127 [1006 to 26132] | 436 [179 to 1061]

6. Primary Outcome: Part C: Maximum Observed Plasma Concentration (Cmax) of M5717
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48, 72, 96, 120, 144, 192, 240, 384, 504, 768 and 1032 hours post-dose
Population: Pharmacokinetic (PK) analysis set included all participants who received M5717,had no clinically important protocol deviations or important events affecting PK, and provide at least one (measurable) post-dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Nanograms per milliliter (ng/mL) | 36.3 (37.0) | 174 (28.7) | 269 (48.2)

7. Primary Outcome: Part C: Time to Reach Maximum Observed Plasma Concentration (Tmax) of M5717
Description: The time to reach the maximum observed plasma concentration (tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 6
Population: Pharmacokinetic (PK) analysis set included all participants who received M5717, had no clinically important protocol deviations or important events affecting PK, and provide at least one (measurable) post-dose concentration.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Hours | 3.75 [1.00 to 12.00] | 2.01 [1.00 to 8.00] | 2.00 [1.50 to 6.02]

8. Primary Outcome: Part C: Terminal Elimination Rate Constant (Lambda z) of M5717
Description: Lambda z determined from the terminal slope of the log-transformed concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: one per hour (1/hour)
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
one per hour (1/hour) | 0.00653 (19.4) | 0.00476 (14.9) | 0.00358 (20.1)

9. Primary Outcome: Part C: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of M5717
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from the determination of the terminal first order (elimination) rate constant (lambda z). AUC0-inf = AUC0-t plus Clast pred/lambda z. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve. Clastpred was the last predicted quantifiable concentration.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Nanogram*hour per milliliter (ng*h/mL) | 3100 (41.0) | 10300 (40.4) | 20000 (37.6)

10. Primary Outcome: Part C: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of M5717
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification (LLOQ), calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
ng*h/mL | 2680 (44.9) | 9470 (42.9) | 19200 (38.9)

11. Primary Outcome: Part C: Area Under the Plasma Concentration-Time Curve From Time Zero to Time 144 Hours After Drug Administration (AUC0-144h) of M5717
Description: The area under the plasma concentration-time curve from time zero to 144 hours after dosing was reported. It is calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48, 72, 96, 120, and 144 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
ng*h/mL | 1930 (34.7) | 6260 (35.1) | 10000 (28.4)

12. Primary Outcome: Part C: Apparent Terminal Half Life (t1/2) of M5717
Description: T1/2 was the time measured for the concentration to decrease by one half. T1/2 was calculated as natural log2 divided by lambda z. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Hours | 106 (19.4) | 146 (14.9) | 193 (20.1)

13. Primary Outcome: Part C: Apparent Total Clearance (CL/f) of M5717
Description: Apparent total body clearance of drug from plasma following extravascular administration, calculated as dose/AUC0-infinity for M5717, whereas AUC0-infinity is area under the plasma concentration-time curve from time zero (dosing time) extrapolated to infinity of unchanged drug calculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-infinity calculated by Clastpred/lambda z, where Clastpred is the predicted plasma concentration at the last sampling time point, calculated from the log linear regression line for lambda z determination at which the measured plasma concentration is at or above lower limit of quantification.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Liter per hour | 38.4 (41.0) | 31.1 (40.4) | 31.9 (37.6)

14. Primary Outcome: Part C: Apparent Volume of Distribution During Terminal Phase (VZ/f) of M5717
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as Vz/f = Dose/(AUC0-infinity multiply by Lambda z) following single dose.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Liter | 5880 (30.1) | 6530 (28.7) | 8890 (26.8)

15. Primary Outcome: Part C: Time Above or Equal to the Predicted M5717 Minimum Inhibitory Concentration (MIC) of 3 ng/mL (t =>3 ng/mL)
Description: Minimal inhibitory concentration (MIC), defined as the concentration at which the relative rate of change in parasitemia is equal to zero.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Hours | 314.55 [213.06 to 392.65] | 518.50 [390.70 to 827.08] | 809.12 [495.92 to 1031.63]

16. Primary Outcome: Part C: Time Above or Equal to the Predicted M5717 Minimum Parasiticidal Concentration (MPC) of 10 ng/mL (t =>10 ng/mL)
Description: Minimal parasiticidal concentration represents the lowest drug concentration value above which parasites decline at a maximal rate.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Hours | 107.47 [36.65 to 139.31] | 281.15 [186.41 to 482.73] | 500.26 [242.97 to 643.18]

17. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of M5717
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng/mL | 7.50 (54.3) | 14.9 (19.7) | 35.7 (41.3) | 146 (37.9) | 267 (25.4) | 642 (53.2) | 988 (40.3) | 1160 (22.7) | 1240

18. Secondary Outcome: Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of M5717
Description: as for outcome 7
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Hours | 1.00 [1.00 to 1.00] | 7.00 [1.00 to 12.00] | 4.00 [0.50 to 8.02] | 3.00 [1.50 to 6.00] | 2.00 [1.00 to 6.00] | 1.75 [1.50 to 10.00] | 1.75 [1.50 to 8.00] | 2.00 [1.50 to 6.00] | 1.50

19. Secondary Outcome: Part A: Terminal Elimination Rate Constant (Lambda z) of M5717
Description: as for outcome 8
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: one per hour (1/hour)
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
one per hour (1/hour) | 0.00523 (39.7) | 0.00523 (29.5) | 0.00478 (28.4) | 0.00447 (17.3) | 0.00382 (25.6) | 0.00411 (38.0) | 0.00386 (16.7) | 0.00383 (31.4) | 0.00493

20. Secondary Outcome: Part A: Apparent Terminal Half Life (t1/2) of M5717
Description: as for outcome 12
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Hours | 133 (39.7) | 133 (29.5) | 145 (28.4) | 155 (17.3) | 181 (25.6) | 169 (38.0) | 180 (16.7) | 181 (31.4) | 140

21. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of M5717
Description: as for outcome 9
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng*h/mL | 997 (23.9) | 1710 (44.3) | 3500 (28.1) | 10100 (24.9) | 17500 (29.7) | 28600 (29.8) | 37800 (28.2) | 52800 (32.4) | 43000

22. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of M5717
Description: as for outcome 10
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng*h/mL | 492 (53.7) | 1250 (50.0) | 2630 (32.6) | 9290 (25.5) | 15800 (40.9) | 27900 (29.7) | 37000 (28.6) | 51300 (33.0) | 42200

23. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero to Time 144 Hours After Drug Administration (AUC0-144h) of M5717
Description: as for outcome 11
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48, 72, 96, 120, and 144 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng*h/mL | 475 (44.0) | 949 (30.3) | 1940 (28.9) | 5830 (29.6) | 9510 (22.4) | 18400 (28.8) | 24200 (24.0) | 32200 (24.8) | 27200

24. Secondary Outcome: Part A: Extrapolated Area Under the Plasma Concentration Curve From Time of Last Quantifiable Sample to Infinity (AUCextra%) of M5717
Description: AUCextra% was calculated as area under the curve from time tlast extrapolated to infinity given as percentage of AUC 0-infinity. Here, tlast is the last sampling time at which the concentration is at or above the lower limit of quantification.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
percentage of AUC0-inf | 45.2 (40.5) | 26.2 (24.3) | 24.0 (25.8) | 6.98 (47.1) | 5.89 (106.5) | 2.36 (33.2) | 2.09 (41.9) | 2.12 (88.7) | 1.78

25. Secondary Outcome: Part A: Apparent Total Clearance (CL/f) of M5717
Description: as for outcome 13
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Liter per hour | 39.9 (23.9) | 46.5 (44.3) | 45.5 (28.1) | 31.7 (24.9) | 27.4 (29.7) | 27.9 (29.8) | 26.3 (28.2) | 27.1 (32.4) | 38.8

26. Secondary Outcome: Part A: Apparent Volume of Distribution During Terminal Phase (VZ/f) of M5717
Description: as for outcome 14
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Liters | 7640 (45.6) | 8890 (18.3) | 9510 (32.9) | 7100 (24.3) | 7160 (24.1) | 6770 (38.7) | 6830 (22.5) | 7060 (24.8) | 7870

27. Secondary Outcome: Part A: Dose Normalized AUC0-inf [AUC(0-inf/Dose)] of M5717
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from the determination of the terminal first order (elimination) rate constant (lambda z). AUC0-inf = AUC0-t plus Clast pred/lambda z. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve. Clastpred was the last predicted quantifiable concentration. Dose normalized was calculated using actual dose, using the formula AUC0-inf/Dose.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng*h/mL/mg | 25.1 (23.9) | 21.5 (44.3) | 22.0 (28.1) | 31.5 (24.9) | 36.5 (29.7) | 35.9 (29.8) | 38.0 (28.2) | 36.9 (32.4) | 25.8

28. Secondary Outcome: Part A: Dose Normalized AUC0-144h [AUC(0-144hour/Dose)] of M5717
Description: The area under the plasma concentration-time curve from time zero to 144 hours after dosing was reported. It is calculated using the mixed log-linear trapezoidal rule (linear up, log down). Dose normalized was calculated using actual dose, using the formula AUC0-144h/Dose.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48, 72, 96, 120, and 144 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng*h/mL/mg | 11.9 (44.0) | 11.9 (30.3) | 12.2 (28.9) | 18.3 (29.6) | 19.9 (22.4) | 23.1 (28.8) | 24.3 (24.0) | 22.5 (24.8) | 16.3

29. Secondary Outcome: Part A: Dose Normalized AUC0-t [AUC( 0-t/Dose)] of M5717
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification (LLOQ), calculated using the mixed log-linear trapezoidal rule (linear up, log down). Dose normalized was calculated using actual dose, using the formula AUC0-t/Dose.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng*h/mL/mg | 12.4 (53.7) | 15.7 (50.0) | 16.5 (32.6) | 29.1 (25.5) | 33.1 (40.9) | 35.0 (29.7) | 37.1 (28.6) | 35.9 (33.0) | 25.3

30. Secondary Outcome: Part A: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M5717
Description: Cmax was obtained directly from the concentration versus time curve. Dose normalized was calculated using actual dose, using the formula Cmax/Dose.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
ng/mL/mg | 0.189 (54.3) | 0.187 (19.7) | 0.224 (41.3) | 0.459 (37.9) | 0.559 (25.4) | 0.805 (53.2) | 0.992 (40.3) | 0.815 (22.7) | 0.743

31. Secondary Outcome: Part A: Time Above or Equal to the Predicted M5717 Minimum Inhibitory Concentration (MIC) of 3 ng/mL (t =>3 ng/mL)
Description: as for outcome 15
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Hours | 84.97 [28.43 to 163.58] | 190.36 [142.93 to 387.46] | 318.49 [266.44 to 439.41] | 551.05 [450.93 to 648.80] | 765.01 [240.48 to 999.95] | 868.99 [542.58 to 944.79] | 832.05 [700.96 to 1031.76] | 1031.17 [647.04 to 1080.71] | 867.02

32. Secondary Outcome: Part A: Time Above or Equal to the Predicted M5717 Minimum Parasiticidal Concentration (MPC) of 10 ng/mL (t=>10 ng/mL)
Description: as for outcome 16
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1
Hours | 0.00 [0.00 to 2.03] | 12.43 [1.40 to 69.80] | 88.02 [46.18 to 159.20] | 272.00 [227.29 to 343.13] | 436.47 [240.32 to 561.56] | 506.34 [312.10 to 548.62] | 531.75 [441.06 to 718.23] | 708.93 [437.26 to 1030.05] | 495.96

33. Secondary Outcome: Part C: Parasite Clearance Time
Description: The parasite clearance time (PCT), defined as the time at which malaria parasite levels decline below detectable levels in blood after treatment, estimated as the time at which the linear portion of the optimal log parasitemia-versus-time relationship intersects the LLOQ concentration line.
Time Frame: Day 1 up to Day 22
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 6 | 7
Hours | 35.8 [31.3 to 40.3] | 54.4 [47.2 to 61.6] | 55.7 [52.9 to 58.5]

34. Secondary Outcome: Part C: Parasite Clearance Half-life (PCT 1/2)
Description: The parasite clearance half-life (PCt1/2), defined as the time needed for parasitemia to be reduced by half during the log-linear phase of parasite clearance, as derived using the slope of the optimal fit of the log-linear relationship of parasitemia decay. It was observed that the decline of parasitemia had a biphasic profile, with the first phase, followed by a second phase (the main clearance phase).
Time Frame: Day 1 up to Day 22
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 6 | 7
Hours
  First Phase | 231.06 [40.93 to NA] — The NA value shown in the upper bound is a stand-in for infinity. | 60.42 [38.63 to 138.6] | 24.66 [20.35 to 31.27]
  Second Phase | 3.52 [3.12 to 4.03] | 3.89 [3.27 to 4.81] | 5.47 [4.78 to 6.41]

35. Secondary Outcome: Part C: Number of Participants With Lag Phase
Description: Lag phase is defined as an initial period after dosing that precedes a steady exponential decline in the parasite count. Lag phase is categorized in lag of 4 hours, lag of 6 hours, lag of 12 hours and lag of 24 hours.
Time Frame: Day 1 to Day 22
Population: Pharmacodynamic (PD) analysis set included all participants who received M5717, had no clinically important protocol deviations or important events affecting PD and provided at least one (measurable) post-dose PD data.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Participants
  Lag of 4 hours | 0 | 6 | 0
  Lag of 6 hours | 3 | 0 | 7
  Lag of 12 hours | 1 | 0 | 0
  Lag of 24 hours | 1 | 0 | 0

36. Secondary Outcome: Part C: Number of Participants With Recrudescence
Description: Recrudescence is as defined as greater than and equal to 5000 blood stage parasites/milliliter (mL) and a 2-fold parasitemia increase within 48 hours, or re-occurrence of malaria symptoms with a malaria clinical score > 6. The malaria clinical score consists of 14 signs/symptoms frequently associated with malaria and graded using a 4-point scale with minimum score is 0 (no symptoms) and the maximum score is 42 (maximum symptoms).
Time Frame: Day 1 to Day 22
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Participants | 3 | 2 | 0

37. Secondary Outcome: Part C: Malarial Clinical Score
Description: The malaria clinical score consists of 14 signs/symptoms frequently associated with malaria and graded using a 4-point scale (absent: 0; mild: 1; moderate: 2; severe: 3) and summed to generate a total malaria clinical score (maximum score possible is 42): headache, myalgia (muscle ache), arthralgia (joint ache), fatigue/lethargy, malaise (general discomfort/uneasiness), chills/shivering/rigors, sweating/hot spells, anorexia, nausea, vomiting, abdominal discomfort, fever, tachycardia and hypotension. Total scores are reported here. The minimum score is 0 (no symptoms) and the maximum score is 42 (maximum symptoms).
Time Frame: Day 1, 2, 3, 4, 5, 6, 7, 9, 11, 13, 15 and 22
Population: Safety Analysis Set included all participants who received investigational medicinal product (M5717 for Part C). Here, Number Analyzed signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Units on a Scale
  Day 1 | 0 (0.4) | 0 (0.0) | 1 (0.8)
  Day 2: number analyzed (Participants) | 6 | 8 | 5
  Day 2 | 0 (0.4) | 1 (0.9) | 0 (0.5)
  Day 3 | 1 (0.8) | 0 (0.5) | 0 (0.5)
  Day 4 | 0 (0.4) | 1 (0.9) | 0 (0.7)
  Day 5 | 0 (0.4) | 0 (0.4) | 0 (0.4)
  Day 6: number analyzed (Participants) | 6 | 2 | 8
  Day 6 | 0 (0.8) | 2 (0.7) | 0 (0.0)
  Day 7: number analyzed (Participants) | 6 | 8 | 1
  Day 7 | 1 (0.5) | 0 (0.5) | 0
  Day 9: number analyzed (Participants) | 6 | 8 | 0
  Day 9 | 0 (0.0) | 0 (0.0) |
  Day 11: number analyzed (Participants) | 6 | 8 | 0
  Day 11 | 0 (0.0) | 0 (0.0) |
  Day 13: number analyzed (Participants) | 0 | 3 | 0
  Day 13 |  | 0 (0.0) |
  Day 15: number analyzed (Participants) | 6 | 8 | 0
  Day 15 | 0 (0.4) | 0 (0.4) |
  Day 22 | 0 (0.0) | 0 (0.0) | 0 (0.0)

38. Secondary Outcome: Part C: Minimum Inhibitory Concentration (MIC) and Minimum Parasiticidal Concentration at 90% (MPC90)
Description: MIC is defined as the minimum concentration of a drug at which parasite counts continue to decrease and is equivalent to equating the rate in the change of parasite to 0. Parasiticidal concentration required for 90% killing (MPC90) is defined as the concentration at which the parasite clearance effect is at 90% of the maximum. The estimated MIC and MPC were derived from the final pharmacodynamics (PD) model and pharmacokinetic (PK)/PD relationship.
Time Frame: Day 1 up to Day 22
Population: as for outcome 35
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
ng/mL
  MIC | 7.59 [2.84 to 20.6] | 7.59 [2.84 to 20.6] | 7.59 [2.84 to 20.6]
  MPC90 | 9.21 [3.45 to 25.0] | 9.21 [3.45 to 25.0] | 9.21 [3.45 to 25.0]

39. Secondary Outcome: Part C: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation of Study Treatment
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered with study drug which does not necessarily had a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 44
Population: Safety Analysis Set included all participants who received investigational medicinal product (M5717 for Part C).
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Participants
  TEAEs | 6 | 8 | 7
  Serious TEAEs | 0 | 0 | 0
  TEAE leading to Discontinuation | 0 | 0 | 0

40. Secondary Outcome: Part C: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Assessments
Description: as for outcome 2
Time Frame: Baseline up to Day 44
Population: Safety Analysis Set included all participants who received investigational medicinal product (M5717 for Part C).
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Participants | 0 | 0 | 0

41. Secondary Outcome: Part C: Number of Participants With Clinically Significant Changes From Baseline in 12-lead Electrocardiograms (ECGs) Findings
Description: The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. Number of participants with clinically significant change from baseline in ECG were reported. Clinical significance was decided by the investigator.
Time Frame: Baseline up to Day 44
Population: Safety Analysis Set included all participants who received investigational medicinal product (M5717 for Part C).
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Participants | 0 | 1 | 1

42. Secondary Outcome: Part C: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate. Number of participants with clinically significant change from baseline in vital signs were reported. Clinical significance was decided by the investigator.
Time Frame: Baseline up to Day 44
Population: Safety Analysis Set included all participants who received investigational medicinal product (M5717 for Part C).
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
Number analyzed (Participants) | 6 | 8 | 8
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For Part A: Baseline up to Day 55. For Part C: Baseline up to Day 44.
Arm/Group | Part A: Placebo (Pooled) | Part A: Cohort 1 SAD: M5717 50 mg | Part A: Cohort 2 SAD: M5717 100 mg | Part A: Cohort 3 SAD: M5717 200 mg | Part A: Cohort 4 SAD: M5717 400 mg | Part A: Cohort 5 SAD: M5717 600 mg | Part A: Cohort 6 SAD: M5717 1000 mg | Part A: Cohort 7 SAD: M5717 1250 mg | Part A: Cohort 8 SAD: M5717 1800 mg | Part A: Cohort 9 SAD: M5717 2100 mg | Part C: M5717 150 mg | Part C: M5717 400 mg | Part C: M5717 800 mg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/1 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/1 | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 13/17 | 6/6 | 5/6 | 3/6 | 4/6 | 3/6 | 4/6 | 5/6 | 6/6 | 1/1 | 6/6 | 8/8 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (Pooled) (N=17) | Part A: Cohort 1 SAD: M5717 50 mg (N=6) | Part A: Cohort 2 SAD: M5717 100 mg (N=6) | Part A: Cohort 3 SAD: M5717 200 mg (N=6) | Part A: Cohort 4 SAD: M5717 400 mg (N=6) | Part A: Cohort 5 SAD: M5717 600 mg (N=6) | Part A: Cohort 6 SAD: M5717 1000 mg (N=6) | Part A: Cohort 7 SAD: M5717 1250 mg (N=6) | Part A: Cohort 8 SAD: M5717 1800 mg (N=6) | Part A: Cohort 9 SAD: M5717 2100 mg (N=1) | Part C: M5717 150 mg (N=6) | Part C: M5717 400 mg (N=8) | Part C: M5717 800 mg (N=8)
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 3
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Catheter site bruise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymph node palpable (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 2 | 1 | 3 | 2 | 1 | 0 | 4 | 0 | 3 | 5 | 4
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03261401/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03261401/SAP_001.pdf